## Postoperative Rehabilitation or Mobilization After Scoliosis Surgery

ID: 2017/53

**Document Date: 02/05/2017** 

## **Study Protocol**

The study was a single-blind randomized clinical trial with parallel group and allocation ratio was 1:1. This study was approved by the Clinical Research Institutional Review Board (No. 2017/53). The study was performed at the Department of Orthopaedics and Traumatology, Turgut Ozal Medical Hospital, Inonu University. Informed written consent was obtained from all participants' parents or legal guardians. The patients who met the inclusion criteria randomly assigned into two groups (Rehabilitation group, Mobilization group) in a ratio of 1:1 through the stratified block randomization method. The patients and the researcher who were responsible for the analyzing of the data were blinded to the randomization results. All data were collected at baseline, 1 week and 6 weeks (only quality of life).

## **Statistical Analysis Plan**

The SPSS (version23; SPSSInc., Chicago, IL, USA) was used to conduct the analysis. Descriptive statistics were presented as mean  $\pm$  standard deviation and percentage. Suitability of variables to normal distribution were analyzed using visual (histogram and probability graphics) and analytical methods (Shapiro-Wilk Test). The differences between both groups were assessed by Chi-squared, Fisher's final test and independent sample t test. Split plot ANOVA was used to compare the pretreatment and posttreatment assessments at baseline, 1 week/6 week in both groups (group: rehabilitation vs mobilization; time: baseline vs 1 week/6 week). VAS, thorax mobility, trunk balance, 2MWT and SRS-22 scales were analyzed for both groups using the split plot ANOVA. A p value of <0.05 was considered to be significant.